CLINICAL TRIAL: NCT05982236
Title: The Psychological and Social Impact of PCOS
Acronym: SPICE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: 2022_0685
Record Dates: First submitted 2023-07-31; First posted 2023-08-08 (Actual); Last update posted 2023-08-25 (Actual); Status verified 2023-08

CONDITIONS: Polycystic Ovary Syndrome
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- PCOS patients
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — Questionnaire on WEPI software (secure data), with link sent by e-mail to patients included in the study, including PCOSQOL, HADS, FACT G7 et ASEX scores.
  Other Names: Questionnaire on WEPI

SUMMARY:
The aim of the study is to assess the association between the quality of life of patients with PCOS and various factors (age, BMI, socio-professional category, delay in diagnostic of PCOS, infertility, hyperandrogenism, parity, history of anxiety and depression, cycles disorders). This study will be proposed to patients known to have PCOS, during a follow-up consultation or a visit to a day hospital in the Gynaecology Department and/or a consultation in the Reproductive Medicine Department. No-objection forms will be collected at the same time. A link will be sent by e-mail to the patient to access the online questionnaire on the WEPI software and complete it after the consultation. Responses to the questionnaire will be collected progressively and stored in a secure RedCAP file.

ELIGIBILITY:
Inclusion Criteria:

* Female sex
* Adult patient (aged 18 or over)
* Able to read and write in French
* diagnosed at a previous consultation as having PCOS according to the Rotterdam criteria (at least 2 out of 3 criteria from:

  * Clinical signs of hyperandrogenism (hirsutism, acne, androgenic alopecia) and/or biochemical signs of hyperandrogenism (total testosterone > 0.39 ng/mL and/or androstenedione > 1.75 ng/mL)
  * Ovulation disorders (infertility, oligomenorrhoea or amenorrhoea or cycle length either <21 days or >35 days),
  * Polymicrocystic ovaries on ultrasound (either 19 or more follicles measuring 2-9 mm in diameter and/or increased ovarian volume (>10 cm3) and/or increased ovarian area (> 5.5 cm²) without presence of cyst or dominant follicle.)
* Informed consent

Exclusion Criteria:

* Patient with no health insurance cover
* Difficulties understanding or speaking French
* Computer (tablet/smartphone) and internet connection required.
* Refusal to take part in research
* Under court protection (guardianship/curatorship/privation of liberty)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with PCOS
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-07-07 (Actual); Primary Completion 2024-04-07 (Estimated); Study Completion 2024-04-07 (Estimated)

PRIMARY OUTCOMES:
Assessment to the The Polycystic Ovary Syndrome Quality of Life scale questionnaire score | Day of inclusion
  according to predefined factors (age, BMI, socio-professional category, delay in diagnosis of Polycystic Ovary Syndrome, infertility, hyperandrogenism, parity, history of anxiety and depression, cycle disorders). Mininum score: 35, maximum score: 245, A higher score means best result

SECONDARY OUTCOMES:
Assessment of the Hospital Anxiety and Depression Scale (HADS) questionnaire score according to predefined factors | Day of inclusion
  minimun: 0 maximum: 42. A higher score means worse result
Assessment of the functional Assessment of Cancer Therapy-General (FACT G7) score according to predefined factors | Day of inclusion
  minimun: 0 maximum: 28 A higher score means worse result
Assessment of the Arizona Sexual Experience Scale (ASEX) score according to predefined factors | Day of inclusion
  minimun: 0 maximum: 30. A higher score means better result

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Lille Hôpital Jeanne de Flandre, Lille, Nord, France

IPD SHARING:
Plan to Share IPD: No